CLINICAL TRIAL: NCT04807790
Title: Effects of "Telerehabılıtatıon Based Structured Home Program Implementatıons" For The Improvement Of Motor Functıon, Activity And Participation In Pre-Schooler Chıldren With Cerebral Palsy
Brief Title: Effects of "Telerehabılıtatıon Based Structured Home Program Implementatıons" Chıldren With Cerebral Palsy
Acronym: (EoTBHPCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mintaze Kerem Gunel, Prof. Doc.Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KA- 20124
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy
Keywords: telerehabilitation; cerebral palsy; home program; participation; activity
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation based structured home program group (Experimental): The structured home program will consist of activities determined by the family members according to the functional level of the child and the activities he / she can not do, and which are determined according to the goals specific to the child. In order to ensure that the structured home program created can be implemented by the family, a 1 hour family training will be provided.
  After the structured home program training, a 45-minute video interview will be held with one of the family members (mother-father-caregiver) once a week, in order to check by the physiotherapist whether the home program is implemented correctly. Video interviews will be the telerehabilitation part of the study.
  Interventions: Other: Telerehabilitation based structured home program applications
- Routine physiotherapy and rehabilitation group (No Intervention): Routine physiotherapy and rehabilitation practices, consist of activities organized by physiotherapists as one or two sessions per week according to the functional levels of children with CP. Routine physiotherapy and rehabilitation applications include increasing postural control, gaining motor development steps, strengthening training, balance training, long-term stretching training, manual therapy, hydrotherapy, hippotherapy and neurodevelopmental therapy approaches.

INTERVENTIONS:
Other: Telerehabilitation based structured home program applications — The structured home program will consist of activities determined by the family members according to the functional level of the child and the activities he / she can not do, and which are determined according to the goals specific to the child. In order to ensure that the structured home program created can be implemented by the family, a 1 hour family training will be provided.
  After the structured home program training, a 45-minute video interview will be held with one of the family members (mother-father-caregiver) once a week, in order to check by the physiotherapist whether the home program is implemented correctly. Video interviews will be the telerehabilitation part of the study.
  Other Names: Routine physiotherapy and rehabilitation group
  Arms: Telerehabilitation based structured home program group

SUMMARY:
The aim of the study is to examine the effectiveness of Telerehabilitation Based Structured Home Program Implementations on functional status, activity and participation in preschool children with Cerebral Palsy.

DETAILED DESCRIPTION:
The structured home program will consist of activities determined by the family members according to the functional level of the child and the activities child can't do, and which are determined according to the goals specific to the child. In order to ensure that the structured home program created can be implemented by the family, a 1 hour family training will be provided.

After the structured home program training, a 45-minute video interview will be held with one of the family members (mother-father-caregiver) once a week, in order to check by the physiotherapist whether the home program is implemented correctly. Video interviews will be the telerehabilitation part of the study.

During routine physiotherapy and rehabilitation practices, activities organized by physiotherapists as one or two sessions per week according to the functional levels of children with CP. Routine physiotherapy and rehabilitation applications include increasing postural control, gaining motor development steps, strengthening training, balance training, long-term stretching training, manual therapy, hydrotherapy, hippotherapy and neurodevelopmental therapy approaches. Telerehabilitation-based structured home program applications, which are given in addition to routine physiotherapy and rehabilitation applications, and only individuals who receive routine physiotherapy and rehabilitation will be followed for 24 weeks. Individuals who receive routine physiotherapy and rehabilitation will be monitored only for control purposes, and a structured home program will be given to the group that receives Telerehabilitation Based Structured Home Program Practices, which are given in addition to routine physiotherapy and rehabilitation applications. The researcher will not be included in the program of the group that only benefits from routine physiotherapy and rehabilitation practices. A total of three evaluations will be made for both groups, after the training before the training and after 12 weeks from the training.

ELIGIBILITY:
Inclusion Criteria:

1. Being in preschool period (3-5 years old)
2. Receiving routine physiotherapy and rehabilitation services 2 sessions in a week
3. Family members being active mobile phone or computer and internet users

Exclusion Criteria:

1. Uncontrolled epileptic seizures
2. Incomplete assesments
3. Family's discontinuation of treatment

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-88 (GMFM-88) | At baseline
  GMFM-66 is a widely used scale to show the improvement in motor function. The KMFM-88 evaluates the motor functional structure in five main positions: supine and prone lying and rolling (A), sitting (B), crawling and kneeling (C), standing (D), walking, running and jumping (E). The highest score is 100, the lowest score is 0.
Quality of Upper Extremity Skills Test (QUEST) | At baseline
  It is used to evaluate the upper extremity motor functions of children. QUEST is a test that evaluates the quality of movement and dexterity of the child with SP. QUEST is concerned with how the child does the activity he or she can do. Examines the quality of upper limb skills in 7 sections. The highest score is 100, the lowest score is 50.

OTHER OUTCOMES:
Segmental Assessment of Trunk Control (SATCO) | At baseline
  It is used to evaluate trunk postural control in children with CP. Examines 7 levels of body control with and without support at C7, T3, T11, L3 and Pelvis level. The highest score is 20, the lowest score is 1.
ABILHAND-KIDS | At baseline
  It evaluates hand skills in children with CP according to the activity frames of ICF-CY. It consists of 21 items. The highest score is 20, the lowest score is 0.
ABILOCO KIDS | At baseline
  It is a scale that evaluates the walking ability of children with CP according to the activity frame of ICF-CY. . 10 maddeden oluşmaktadır. The highest score is 20, the lowest score is 0.
Goal Attainment Scale (GAS) | At baseline
  It is used to evaluate the effect of individualized, goal directed physiotherapy and rehabilitation programs for children with CP. In order to measure the effect of the treatment, specific goals for the child are determined together with the family, child and experts. Goals; It is graded at five levels, from -2 to 2.
LIFE-H | At baseline
  It has been developed to evaluate the participation in life of children with CP. It consists of 11 sub-headings: nutrition, physical fitness, personal care, mobility, interpersonal communication, social roles, education, recreational activities, responsibilities, housing, and social life. The highest score is 10, the lowest score is 0.
Canadian Occupational Performance Measure | At baseline
  It is used to evaluate activity performance and satisfaction levels in individuals. This assessment scale is a measure that determines the problems faced by individuals in the field of activity performance through a semi-structured interview. This measurement evaluates the activity performance problems of individuals with the performance and satisfaction scores they give themselves. The highest score is 10, the lowest score is 0.
Europian Child Environment Questionnaire ECEQ | At baseline
  It was created in order to evaluate the environmental factors in children with CP and to determine the needs and accessibility to the needs. It is a valid (ICC> 0.95) scale consisting of 60 questions that evaluate the conditions in home, school and social life under three main sub-headings: physical environment, social support and attitudes. Scored "0: Not required", "1: Necessary and mostly accessible", "2: Required but mostly unavailable" to determine need and availability.
Compliance of Parents of Children with Cerebral Palsy to Home Program Questionairre (CPHP-Q) | At baseline
  It is a scale that examines the reasons for parents with children with CP between the ages of 2 and 18 not to adapt to the home program within the scope of personal and environmental factors. Scale items were created under the umbrella of ICF-CY frame. It has proven to be highly valid and reliable. It consists of 22 items. The highest score is 110, the lowest score is 22.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sel SA, Gunel MK, Erdem S, Tuncdemir M. Effects of Telerehabilitation-Based Structured Home Program on Activity, Participation and Goal Achievement in Preschool Children with Cerebral Palsy: A Triple-Blinded Randomized Controlled Trial. Children (Basel). 2023 Feb 22;10(3):424. doi: 10.3390/children10030424. PMID 36979982